CLINICAL TRIAL: NCT00049010
Title: Prospective Study of Melastatin Expression in Predicting the Risk for Developing Local Regional Metastases of Primary Melanoma
Brief Title: Diagnostic Study to Predict the Risk of Developing Metastatic Cancer in Patients With Stage I or Stage II Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Purpose: Diagnostic
Other Study IDs: CALGB-500105; U10CA031946 (NIH); CALGB-500105; CDR0000257230 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Melanoma (Skin)
Keywords: stage I melanoma; stage II melanoma
MeSH Terms: conditions — Melanoma | interventions — Comparative Genomic Hybridization; Cytogenetic Analysis; In Situ Hybridization, Fluorescence; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group 1 (Experimental): Melastatin mRNA expression is determined by in situ hybridization using tissue from primary tumor and lymph nodes. Tissue is also examined by immunohistochemical staining using antibodies to S-100 and MART-1. Patients do not receive the results of these tests nor do the results influence individual therapy.
  Patients are followed every 4 months for 3.5 years.
  Interventions: Genetic: comparative genomic hybridization; Genetic: cytogenetic analysis; Genetic: fluorescence in situ hybridization; Other: immunohistochemistry staining method

INTERVENTIONS:
Genetic: comparative genomic hybridization
Genetic: cytogenetic analysis
Genetic: fluorescence in situ hybridization
Other: immunohistochemistry staining method

SUMMARY:
RATIONALE: Diagnostic procedures that analyze surgically-removed tumor tissue and lymph node samples may help doctors identify patients with melanoma who are at risk for developing metastatic cancer.

PURPOSE: This clinical trial is studying tumor tissue and lymph node samples to see how well they work in predicting the development of metastatic cancer in patients with stage I or stage II melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Correlate degree of melastatin gene expression with risk of developing local regional metastases in patients with primary stage I or II melanoma.
* Correlate melastatin expression prospectively with event-free survival of these patients.

OUTLINE: This is a multicenter study.

Melastatin mRNA expression is determined by in situ hybridization using tissue from primary tumor and lymph nodes. Tissue is also examined by immunohistochemical staining using antibodies to S-100 and MART-1. Patients do not receive the results of these tests nor do the results influence individual therapy.

Patients are followed every 4 months for 3.5 years.

PROJECTED ACCRUAL: A total of 300 patients will be accrued for this study within 3.5 years.

ELIGIBILITY:
1. Histologically documented primary AJCC stage I or II melanoma. Evidence of ulceration, vertical growth phase, regression, lymphocytic infiltration, vascular invasion, microscopic satellitosis, and mitotic rate shall be noted.
2. Patients planning to undergo a sentinel lymph node biopsy, or an elective lymph node dissection of an anatomic draining region from the index primary melanoma.
3. ≥18 years of age
4. Patients must be registered prior to planned surgery. The surgery must be performed within 45 days following registration.
5. No concurrent active malignancy other than carcinoma in situ of the cervix and basal cell carcinoma of the skin, or history of any other primary malignancy including previously primary melanoma.
6. Tissue blocks: one of primary tumor tissue taken from region of greatest Breslow thickness. Note: If blocks cannot be sent due to institutional policy, slides may be substituted for the locks per the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2002-09; Primary Completion 2006-03 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival | Up to 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: F. Stephen Hodi, MD, Study Chair — Dana-Farber Cancer Institute
Locations (27):
- United States (27):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Commonwealth Hematology-Oncology P.C. - Worcester, Worcester, Massachusetts
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Capital Region Cancer Center, Jefferson City, Missouri
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - CCOP - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - Community General Hospital of Greater Syracuse, Syracuse, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital at Lifespan, Providence, Rhode Island
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia